CLINICAL TRIAL: NCT07182071
Title: Feasibility of a 10-Week Physical Activity Program for Mothers of Children With Developmental Disabilities
Brief Title: 10-Week Physical Activity Program for Mothers of Children With Developmental Disabilities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0981; Protocol Version 7/9/2025 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2025-09-16; First posted 2025-09-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Caregiver Burden
Keywords: mothers; autism; down syndrome; disabilities; fitness
MeSH Terms: conditions — Caregiver Burden; Autistic Disorder; Down Syndrome | interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Program (Experimental): This group will enroll in the 10-week program immediately.
  Interventions: Behavioral: Physical Activity Program
- Waitlist Control (Active Comparator): This group will enroll and then be offered the 10-week program next year.
  Interventions: Behavioral: Waitlist for Physical Activity Program

INTERVENTIONS:
Behavioral: Physical Activity Program — Three 60-minute supervised group exercise sessions per week for 10 weeks, led by a certified instructor.
  Arms: Physical Activity Program
Behavioral: Waitlist for Physical Activity Program — Three 60-minute supervised group exercise sessions per week for 10 weeks, led by a certified instructor.
  Arms: Waitlist Control

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of a 10-week supervised Physical Activity program for mothers of children with developmental disabilities. 30 participants will be enrolled: 15 into an Intervention group and 15 into a Waitlist Control group.

DETAILED DESCRIPTION:
The specific aims of this study are:

* Aim 1: Determine the feasibility and acceptability of a 10-week supervised resistance training program for mothers of autistic children.
* Aim 2: Determine the potential health benefits of the 10-week physical activity program on psychological and physical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Be a mother of a child with a diagnosed developmental disability (e.g., autism spectrum disorder, Down syndrome, intellectual disability) ages 4-11.
* Be able to engage in moderate-intensity exercise three times per week.
* Be able to walk independently for at least a quarter of a mile without assistance.
* Have reliable childcare arrangements during program sessions (please note: childcare will not be provided).
* Be available and willing to attend scheduled assessments and group sessions throughout the 10-week program.

Exclusion Criteria:

* Are currently pregnant.
* Have a physical disability or medical condition that prevents safe participation in physical activity.
* Are already engaged in physical activity programs more than twice per week.
* Have diagnosed mental health conditions that may interfere with consistent attendance or the ability to provide informed consent.
* Are unable to communicate effectively in English.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | through enrollment (up to 12 weeks)
Feasibility: Percent of Sessions Attended | up to 12 weeks
Feasibility: Number of Participants Who Complete the study | up to 12 weeks
Acceptability: Participant Experiences | up to 12 weeks
  Measured qualitatively via semi-structured post-intervention interviews, summarized and reported by participant count.
Acceptability: Participant Satisfaction | up to 12 weeks
  Measured qualitatively via semi-structured post-intervention interviews, summarized and reported by participant count.
Acceptability: Challenges to Participation | up to 12 weeks
  Measured qualitatively via semi-structured post-intervention interviews, summarized and reported by participant count.
Acceptability: Facilitators to Participation | up to 12 weeks
  Measured qualitatively via semi-structured post-intervention interviews, summarized and reported by participant count.

SECONDARY OUTCOMES:
Efficacy: Grip Strength | baseline, week 5, week 10
  The participant will squeeze a handheld dynamometer as hard as possible to measure hand and forearm strength, recorded in kilograms.
Efficacy: Number of Push-Ups Participant Completes with Proper Form | baseline, week 5, week 10
  The participant will perform as many push-ups as possible with proper form to test upper-body endurance.
Efficacy: Five Times Sit to Stand Test (FTSST) | baseline, week 5, week 10
  The amount of time it takes for a participant to transfer from seated to standing and back to sitting five times.
Efficacy: Percent Body Fat and Lean Mass | baseline, week 5, week 10
  Body composition is measured via Bioelectrical Impedance Analysis (BIA). The participant will stand barefoot on a bioelectrical impedance device to estimate body fat and muscle levels.
Efficacy: Fat Mass and Fat-Free Mass in Kilograms | baseline, week 5, week 10
  Body composition is measured via Bioelectrical Impedance Analysis (BIA). The participant will stand barefoot on a bioelectrical impedance device to estimate body fat and muscle levels.
Generalized Anxiety Disorder-7 (GAD-7) | baseline, week 5, week 10
  Scored from 0-21 where higher scores indicate increased anxiety.
Perceived Stress Scale (PSS) | baseline, week 5, week 10
  Scored from 0-40 where higher scores indicate increased stress.
Patient Health Questionnaire-8 (PHQ-8) | baseline, week 5, week 10
  Scored from 0-24 where higher scores indicate increased symptoms of depression
Penn State Worry Questionnaire (PSWQ) | baseline, week 5, week 10
  Scored from 16-80 where higher scores indicate increased worry.
SF-12 Health Survey | baseline, week 5, week 10
  Perceived physical and mental health subscales each scored from 0-100 with higher scores indicating better perceived physical and mental health.
International Physical Activity Questionnaire (IPAQ) | baseline, week 5, week 10
  The IPAQ assesses physical activity during the previous 7 days by asking participants how many days and how many minutes per day they engaged in vigorous activity, moderate activity, walking, and sitting. The responses are converted into metabolic equivalent (MET) minutes per week by multiplying the minutes of activity per week by an assigned MET value (walking = 3.3 METs, moderate activity = 4.0 METs, vigorous activity = 8.0 METs). The total physical activity score is the sum of MET-minutes/week across the activity categories. Higher scores reflect greater levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, PhD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No